CLINICAL TRIAL: NCT04806633
Title: Dapagliflozin to Prevent the Incidence of Contrast Induced Nephropathy After Heart Catheterization and Percutaneous Coronary Intervention
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Professor, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2663
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Left Cardiac Catheterization; Percutaneous Coronary Intervention; Acute Kidney Injury; Sodium-glucose Co-transporter 2 Inhibitors
Keywords: dapaglifozin; iodinated contrast media; Sodium-glucose Co-transporter 2 Inhibitors; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): Patients who will be randomized to receive dapagliflozin following cardiac catheterization and PCI
  Interventions: Drug: Dapagliflozin 5mg
- Placebo (Placebo Comparator): Patients who will be randomized to receive placebo following cardiac catheterization and PCI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 5mg — Patients randomized in this arm will receive dapagliflozin at a dose of 5mg once daily.
  Arms: Dapagliflozin
Drug: Placebo — Patients randomized in this arm will receive placebo.
  Arms: Placebo

SUMMARY:
Left heart catheterization and percutaneous coronary intervention (PCI) has become a useful tool in interventional cardiology, in which iodinated contrast media is used. Although the use of iodinated contrast media (CM) is considered to be safe in patients with normal renal function, it is risky in patients with known chronic renal insufficiency (CKD) and diabetes mellitus. Contrast induced nephropathy (CIN) remains one of the most leading causes of in hospital acute kidney injury (AKI), affecting morbidity and mortality. There are various mechanisms through which CM develop their nephrotoxic effects, including renal vasoconstriction and medullary hypoxia, tubular cell toxicity and reactive oxygen species formation.

Inhibitors of type 2 sodium- glucose co-transporter (SGLT2i) is a relatively recent addition to the array of anti-diabetic agents, becoming part of everyday clinical practice. However, although SGLT2i were first used solely as antidiabetics because of their glycosuric effect, further research demonstrated that these drugs may independently reduce cardiovascular events, especially in patients with heart failure, a benefit that was consistent among diabetic and non-diabetic patients. Moreover, pleiotropic effects have been observed, including a reno-protective action. In addition to the effects mediated by intrarenal hemodynamic changes, SGLT2-i also have direct anti-inflammatory and antifibrotic nephroprotective effects. Indeed, SGLT2-i suppress the production of reactive oxygen species, lessening glomerulosclerosis and tubulo-interstitial fibrosis.

These findings suggest that the use of SGLT2i could offer benefit by reducing/ preventing the nephrotoxic effects of contrast media leading to the assumption that the use of these drugs could prevent the incidence nephropathy after cardiac catheterization and percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Written informed consent
* Glomerular Filtration Rate (GFR)≥ 30 ml/min/1.73m2 [CKD stage G1-G3]
* Percutaneous coronary intervention in patients with NSTEMI, UA, STCD and asymptomatic patients

Exclusion Criteria:

* Active malignancy
* Participation in other intervention study
* Class I or equivalent indication for treatment with a SGLT2 inhibitor
* Pregnancy or willing of pregnancy during the follow up period
* Active urogenital infection
* Diabetes mellitus type 1
* History of diabetic ketoacidosis
* Cardiogenic shock
* eGFR < 29 ml/min/1.73m2

  * Patients with an indication for SGLT2 inhibitor will be included in a prospective registry. Their treatment will be determined by their attending physicians.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1722 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of incidence of acute kidney injury (AKI) between the two study arms | 1 month
  AKI is defined defined as an absolute creatinine level increase of at least 0.3 mg/dL (≥26.5 μmol/L) or at least 1.5-fold from baseline.

SECONDARY OUTCOMES:
Development of at least Stage 2 AKI (according to the KDIGO criteria), i.e. Increase in sCR>2.0-fold from baseline. | 1 month

OTHER OUTCOMES:
Incidence (cases per 100 patient-years) of hypoglycemia in both arms Any episode of hypoglycemia defined as serum glucose 60< mg/dl associated with symptoms of hypoglycemia. | 1 month
Incidence (cases per 100 patient-years)of diabetic ketoacidosis. | 1 month
  Any episode of metabolic acidosis (pH<7.3) with decreased serum bicarbonate (<18mEq/ml) and
Incidence (cases per 100 patient-years)of lower urinary tract infections | 1 month
Comparison of all cause mortality between the two groups | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Deftereos, Prof., Principal Investigator — 2nd Department of Cardiology, National and Kapodistrian University of Athens, Faculty of Medicine, Athens, Greece
Locations (2):
- Greece (2):
  - Cardiology Department, Athens General Hospital "G. Gennimatas", Athens
  - 2nd Department of Cardiology, National and Kapodistrian University of Athens, Faculty of Medicine, Athens, Greece., Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aurelio A, Durante A. Contrast-induced nephropathy in percutaneous coronary interventions: pathogenesis, risk factors, outcome, prevention and treatment. Cardiology. 2014;128(1):62-72. doi: 10.1159/000358042. Epub 2014 Feb 18. PMID 24557146
- [Result] Garofalo C, Borrelli S, Liberti ME, Andreucci M, Conte G, Minutolo R, Provenzano M, De Nicola L. SGLT2 Inhibitors: Nephroprotective Efficacy and Side Effects. Medicina (Kaunas). 2019 Jun 11;55(6):268. doi: 10.3390/medicina55060268. PMID 31212638
- [Result] McCullough PA, Choi JP, Feghali GA, Schussler JM, Stoler RM, Vallabahn RC, Mehta A. Contrast-Induced Acute Kidney Injury. J Am Coll Cardiol. 2016 Sep 27;68(13):1465-1473. doi: 10.1016/j.jacc.2016.05.099. PMID 27659469
- [Result] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Result] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Result] Ishibashi Y, Matsui T, Yamagishi S. Tofogliflozin, A Highly Selective Inhibitor of SGLT2 Blocks Proinflammatory and Proapoptotic Effects of Glucose Overload on Proximal Tubular Cells Partly by Suppressing Oxidative Stress Generation. Horm Metab Res. 2016 Mar;48(3):191-5. doi: 10.1055/s-0035-1555791. Epub 2015 Jul 9. PMID 26158396
- [Result] Fioretto P, Zambon A, Rossato M, Busetto L, Vettor R. SGLT2 Inhibitors and the Diabetic Kidney. Diabetes Care. 2016 Aug;39 Suppl 2:S165-71. doi: 10.2337/dcS15-3006. PMID 27440829